CLINICAL TRIAL: NCT01610518
Title: The Glycemic Response Elicited by Beta-glucans of Different Physical Properties and Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guelph Food Research Centre (Other Government)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. Susan M. Tosh, Research Scientist, Guelph Food Research Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UT25964
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: postprandial blood glucose; dietary fiber; beta-glucan
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — beta-glucan, (1-3)(1-4)-

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- 250 mL medium viscosity (Experimental): 250 mL beverage containing 4g low molecular weight oat beta-glucan and 50g glucose
  Interventions: Dietary Supplement: oat beta-glucan
- 600 mL low viscosity (Experimental): 600 mL beverage containing 4g low molecular weight oat beta-glucan and 50g glucose
  Interventions: Dietary Supplement: oat beta-glucan
- 250 mL high viscosity (Experimental): 250 mL beverage containing 4g high molecular weight oat beta-glucan and 50g glucose
  Interventions: Dietary Supplement: oat beta-glucan
- 600 mL medium viscosity (Experimental): 600 mL beverage containing 4g high molecular weight oat beta-glucan and 50g glucose
  Interventions: Dietary Supplement: oat beta-glucan
- 250mL control (Placebo Comparator): 250 mL beverage containing 50g glucose
  Interventions: Dietary Supplement: Placebo
- 600mL control (Placebo Comparator): 600mL beverage containing 50g glucose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: oat beta-glucan — 4g dose for each arm of trial. Form (volume and viscosity) varies between arms. 2h acute trial beginning between 8 and 10 am. Minimum 1 day wash out between arms.
  Other Names: oat soluble fibre
  Arms: 250 mL high viscosity; 250 mL medium viscosity; 600 mL low viscosity; 600 mL medium viscosity
Dietary Supplement: Placebo — Control without beta-glucan. Form (volume) varies between arms. 2h acute trial beginning between 8 and 10 am. Minimum 1 day wash out between arms.
  Arms: 250mL control; 600mL control

SUMMARY:
The ability of oat β-glucan to lower postprandial glycemic responses has been attributed to the viscosity of the solution in which the fibre is solubilized. To our knowledge, no studies have investigated the effect of β-glucan solutions on glycemic response when concentration, and thus viscosity, is varied by changing the solution volume but not the β-glucan dose. Therefore, the investigators will test the effects of altering β-glucan solution viscosity by altering solution volume at a fixed amount of β-glucan fibre.

DETAILED DESCRIPTION:
The ability of β-glucan to lower postprandial glycemic responses has been attributed to the viscosity of the solution in which the fibre is solubilized. It has been demonstrated that the viscosity of a β-glucan solution increases with the molecular weight (MW) of β-glucan polymers, as well as the dose or concentration (C) of those polymers in solution. Numerous studies have shown that glycemic response-lowering is strengthened when the C of a β-glucan solution of fixed liquid volume is increased by increasing β-glucan dose. However, the C of a β-glucan solution depends on not only the amount of fibre present but also on the solution volume. To our knowledge, no studies have investigated the effect of β-glucan solutions on glycemic response when C, and thus viscosity, is varied by changing the solution volume but not the β-glucan dose. Therefore, the investigators will test the effects of altering β-glucan solution viscosity by altering solution volume at a fixed amount of β-glucan fibre. Knowing how to incorporate β-glucan into solution so that its physiological benefits are preserved will assist in the development of β-glucan-containing functional foods.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women

Exclusion Criteria:

* BMI greater than or equal to 35
* known to have diabetes, HIV, hepatitis or a heart condition
* use of medications or having a condition which may harm the subjects
* use of medication which may affect the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
postprandial blood glucose | 2 h
  Two fasting blood samples spaced 5 minutes apart (-5 min and 0 min) were collected by finger-prick using a monoejector lancet device. Immediately following the collection of the second blood sample, subjects consumed a test solution and 250mL of a beverage of their choice (water, tea or coffee with milk and/ or artificial sweetener aspartame). Subjects received the same beverage and volume of that beverage for each test in the study. Additional finger-prick blood samples were taken at 10, 20, 30, 40, 50, 60, 90 and 120 minutes after the start of the meal.

CONTACTS AND LOCATIONS:
Locations (1):
- GILabs, Toronto, Ontario, Canada

REFERENCES:
- [Background] Wolever TM, Jenkins DJ, Jenkins AL, Josse RG. The glycemic index: methodology and clinical implications. Am J Clin Nutr. 1991 Nov;54(5):846-54. doi: 10.1093/ajcn/54.5.846. PMID 1951155
- [Background] Wood PJ, Beer MU, Butler G. Evaluation of role of concentration and molecular weight of oat beta-glucan in determining effect of viscosity on plasma glucose and insulin following an oral glucose load. Br J Nutr. 2000 Jul;84(1):19-23. PMID 10961156